CLINICAL TRIAL: NCT04334824
Title: Use of Hydrochlorothiazide and the Risk of Skin Cancer
Brief Title: Hydrochlorothiazide and Risk of Skin Cancer
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q19-05
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-06

CONDITIONS: Non-melanoma Skin Cancer; Melanoma; Hypertension
Keywords: Non-melanoma Skin Cancer; Melanoma; Hydrochlorothiazide; Hypertension
MeSH Terms: conditions — Melanoma; Hypertension | interventions — Hydrochlorothiazide; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hydrochlorothiazide: Patients who received a new prescription for hydrochlorothiazide (alone or in combination with non-ACE inhibitor antihypertensive drugs) at cohort entry, and did not have a previous prescription for any antihypertensive drug any time before cohort entry.
  Interventions: Drug: Hydrochlorothiazide
- Angiotensin-converting enzyme (ACE) inhibitors: Patients who received a new prescription for an ACE inhibitor (alone or in combination with non-hydrochlorothiazide antihypertensive drugs) at cohort entry, and did not have a previous prescription for any antihypertensive drug any time before cohort entry.
  Interventions: Drug: Angiotensin-converting enzyme (ACE) inhibitors

INTERVENTIONS:
Drug: Hydrochlorothiazide — Exposure to hydrochlorothiazide will be defined as a prescription for hydrochlorothiazide alone or in combination with non-ACE inhibitor antihypertensive drugs at cohort entry date.
  Other Names: ATC C03AA03
  Groups: Hydrochlorothiazide
Drug: Angiotensin-converting enzyme (ACE) inhibitors — Exposure to ACE inhibitors will be defined as a prescription for an ACE inhibitor alone or in combination with non-hydrochlorothiazide antihypertensive drugs at cohort entry date.
  Other Names: ATC C09A, C09B
  Groups: Angiotensin-converting enzyme (ACE) inhibitors

SUMMARY:
The purpose of this study is to determine whether the use of hydrochlorothiazide is associated with an increased risk of skin cancer compared with the use of angiotensin-converting enzyme (ACE) inhibitors. More specifically, the investigators will assess the risk of non-melanoma and melanoma skin cancer. The investigators hypothesize that the use of hydrochlorothiazide is associated with an increased risk of skin cancer compared with ACE inhibitors.

The investigators will carry out separate population-based cohort studies using administrative health databases from seven Canadian provinces and the United States. The study cohort will be defined by the initiation of hydrochlorothiazide or an ACE inhibitor, with follow-up until an incident diagnosis of non-melanoma or melanoma skin cancer. The results from the separate sites will be combined to provide an overall assessment of the risk of non-melanoma and melanoma skin cancer in users of hydrochlorothiazide.

DETAILED DESCRIPTION:
The study objective is to determine whether the use of hydrochlorothiazide is associated with an increased risk of skin cancer compared with the use of angiotensin-converting enzyme (ACE) inhibitors. More specifically, the investigators will assess whether hydrochlorothiazide is associated with the risk of non-melanoma and melanoma skin cancer.

A common-protocol approach will be used to conduct retrospective cohort studies using administrative health data from seven Canadian provinces (Alberta, British Columbia, Manitoba, Nova Scotia, Ontario, Quebec, and Saskatchewan) and the United States (US) MarketScan database. Briefly, the Canadian databases include population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs. Prescription drug data are limited to those aged 65 years old and older in Alberta, Nova Scotia, and Ontario. The US MarketScan database includes individuals and their dependents covered by large US employer health insurance plans, and government and public organizations.

A standardized mortality ratio weighted cohort analysis will be conducted. In each jurisdiction, the investigators will assemble a study cohort that includes all patients aged 40 years or older (or 66 years or older in Alberta, Nova Scotia, and Ontario) newly-treated with hydrochlorothiazide or an ACE inhibitor between April 1, 1995 and March 31, 2018 (or the latest date of data availability at each site). The date of study cohort entry will be defined by the dispensation date of the newly prescribed hydrochlorothiazide or ACE inhibitor. Patients will be followed starting 366 days after study cohort entry until an incident diagnosis of non-melanoma or melanoma, or censored upon switching to a study drug, death, end of coverage or end of the study period (March 31, 2018), whichever occurs first.

Exposure will be defined as a prescription for hydrochlorothiazide or an ACE inhibitor on the date of cohort entry. The exposures will be lagged by one year in order to consider a minimum cancer latency period between treatment initiation and the diagnosis of skin cancer. Analyses will be conducted using a modified intention-to-treat approach. The outcomes of interest will be non-melanoma and melanoma skin cancer.

Weighted Cox proportional hazards models with calendar year as a strata will be used to estimate site-specific adjusted hazard ratios (HR) and corresponding 95% confidence intervals (CI) for each outcome of interest among hydrochlorothiazide users compared to ACE inhibitor users. In order to reflect the Canadian context, the primary analysis will be restricted to Canadian data and the US MarketScan data will be used only in a secondary analysis. Secondary analyses will be conducted for each outcome of interest. These will include the following: 1) as-treated, 2) cumulative duration of use, 3) dose-response relation, 4) effect modification by age (≤65, 66-74, and ≥75 years), sex and immunosuppressive status, and 5) time since initiation of treatment (<3, 3-5, and >5 years). For non-melanoma, events will be further classified into basal cell carcinoma or squamous cell carcinoma sub-types in jurisdictions where data is available. Four sensitivity analyses will be performed to assess the robustness of study results and address some of the study limitations. Site-specific results from the Canadian sites will be combined by random-effects meta-analysis to provide an overall assessment of the risk of non-melanoma and melanoma skin cancer in hydrochlorothiazide users compared to ACE inhibitor users. Four additional analyses at the meta-analysis level will be conducted. These will include the following: 1) using fixed-effects model, 2) pooling results only from jurisdictions where non-melanoma sub-type differentiation is available, 3) pooling results from all sites including the US MarketScan data, and 4) pooling results by jurisdictions with and without cancer registry data.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years or older (or 66 years or older in Alberta, Nova Scotia and Ontario) newly-treated with hydrochlorothiazide or an ACE inhibitor between April 1, 1995 and March 31, 2018 (or the latest date of data availability at each site)

Exclusion Criteria:

* Patients with less than one year of health coverage before cohort entry
* Patients with a previous prescription of any antihypertensive drug at any time before cohort entry
* Patients with a diagnosis of any type of skin cancer (non-melanoma and melanoma) at any time before cohort entry
* Patients with a diagnosis of HIV at any time before cohort entry
* Patients with a history of solid organ transplant at any time before cohort entry
* Patients with less than one year of follow-up after cohort entry

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, the investigators will assemble a study cohort that includes all patients aged 40 years or older newly-treated with hydrochlorothiazide or an ACE inhibitor between April 1, 1995 and March 31, 2018 (or the latest date of data availability at each site). The date of study cohort entry will be defined by the dispensation date of the newly prescribed hydrochlorothiazide or ACE inhibitor.
Sampling Method: Probability Sample
Enrollment: 2953748 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Non-melanoma skin cancer | Patients will be followed starting 366 days after study cohort entry until an incident diagnosis of non-melanoma skin cancer, censoring or for up to 275 months, whichever occurs first.
  Incident non-melanoma skin cancer events will be identified using either cancer registry information (where available), or defined using an algorithm adapted from Chan et al., 2016. An event will be defined by the presence of a diagnosis code for non-melanoma skin cancer (ICD-9: 173.x; ICD-10: C44.x) plus a procedure code in hospital or physician claims data.
Melanoma skin cancer | Patients will be followed starting 366 days after study cohort entry until an incident diagnosis of melanoma skin cancer, censoring or for up to 275 months, whichever occurs first.
  Incident melanoma skin cancer events will be identified using either cancer registry information (where available), or defined using an algorithm. An event will be defined by the presence of a diagnosis code for malignant melanoma (ICD-9: 172.x; ICD-10: C43.x) plus a procedure code in hospital or physician claims data.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Azoulay, PhD, Principal Investigator — Centre for Clinical Epidemiology, Lady Davis Institute, Jewish General Hospital
Locations (1):
- Centre for Clinical Epidemiology, Lady Davis Institute, Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan AW, Fung K, Tran JM, Kitchen J, Austin PC, Weinstock MA, Rochon PA. Application of Recursive Partitioning to Derive and Validate a Claims-Based Algorithm for Identifying Keratinocyte Carcinoma (Nonmelanoma Skin Cancer). JAMA Dermatol. 2016 Oct 1;152(10):1122-1127. doi: 10.1001/jamadermatol.2016.2609. PMID 27533718
- [Background] Azoulay L, St-Jean A, Dahl M, Quail J, Aibibula W, Brophy JM, Chan AW, Bresee L, Carney G, Eltonsy S, Tamim H, Paterson JM, Platt RW; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Hydrochlorothiazide use and risk of keratinocyte carcinoma and melanoma: A multisite population-based cohort study. J Am Acad Dermatol. 2023 Aug;89(2):243-253. doi: 10.1016/j.jaad.2023.04.035. Epub 2023 Apr 25. PMID 37105517
- See also: This is the website describing the general functions of the organization, other CNODES projects, and investigator profiles. — http://www.cnodes.ca